CLINICAL TRIAL: NCT07167394
Title: The Effect of Presenting Restorative Dental Treatments in a Game Format Using Virtual Reality Glasses on Anxiety and Pain Perception in Children
Brief Title: The Effect of Virtual Reality Glasses on Pain Perception
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Levent Özer, professor, Ankara University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023.18/2
Record Dates: First submitted 2025-07-08; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Virtual Reality; Dental Anxiety
Keywords: virtual reality; dental anxiety; dental pain; behavior management
MeSH Terms: conditions — Toothache

STUDY DESIGN:
Intervention Model Description: The study consist of two arms including Virtual Reality Game Group and Tell-Show-Do Group.
Who Masked: Outcomes Assessor
Masking Description: Although the intervention is not blinded to participants or care providers due to the visible nature of the VR headset and behavioral techniques, the individuals evaluating outcome measures (such as anxiety and pain scores) are blinded to group assignment. Self-reported scales are collected by an independent researcher not involved in the intervention delivery. Additionally, the data analysis will be conducted using anonymized group labels (Arm 1 / Arm 2), ensuring that the statistician remains blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Virtual Reality Game Group (Experimental): Children in this group will receive restorative dental treatment following a virtual reality-based animated educational game presented via VR headset. The game introduces each treatment step in a child-friendly narrative to reduce anxiety and perceived pain.
  Interventions: Procedure: Interactive Virtual Reality Guidance with Restorative Dental Treatment
- Tell-Show-Do Group (Experimental): Children in this group will receive the same restorative dental treatment after conventional behavioral preparation using the Tell-Show-Do technique, where each procedure is verbally explained and visually demonstrated prior to treatment.
  Interventions: Procedure: Tell-Show-Do Guidance with Restorative Dental Treatment

INTERVENTIONS:
Procedure: Interactive Virtual Reality Guidance with Restorative Dental Treatment — Participants in this group will undergo a standardized restorative dental procedure on mandibular primary molars involving local anesthesia, caries excavation, and compomer restoration. Prior to the treatment, children will wear a virtual reality (VR) headset through which they will experience an interactive, animated educational game.
  The VR content simulates the treatment steps-including sitting in the chair, receiving local anesthesia, caries removal, filling, and polishing-using engaging characters and storytelling. The aim is to reduce anxiety and perceived pain through immersive visual and cognitive distraction while standard dental procedures are being performed.
  Arms: Virtual Reality Game Group
Procedure: Tell-Show-Do Guidance with Restorative Dental Treatment — Participants in this group will also receive a standardized restorative dental procedure identical to the VR group, including local anesthesia, caries removal, and compomer filling of mandibular primary molars. Behavioral preparation will be conducted using the conventional Tell-Show-Do technique. The clinician will verbally explain each step, demonstrate the procedure using visual and tactile tools in a child-friendly manner, and then proceed with the actual intervention. This method aims to reduce dental fear and increase compliance by familiarizing the child with the clinical environment before the surgical procedure.
  Arms: Tell-Show-Do Group

SUMMARY:
Positive experiences during a child's first dental visit contribute to the development of both acute and long-term positive attitudes toward dentists and dental treatments. However, some children may find dental visits stressful or frightening due to several factors, including being in an unfamiliar environment, fear of pain, negative remarks about dentists they might have heard from others, the sounds of dental equipment, bright lights, or even their parents' anxious demeanor. Addressing these fears and implementing strategies to reduce anxiety and alter pain perception can make dental visits smoother. Such measures also positively influence children's oral health, dental development, future dental experiences, eating habits, general health, and self-confidence.

On the contrary, if the first dental experience is associated with pain and anxiety, this can condition children-particularly those who are more sensitive-to develop persistent dental anxiety. In severe cases, repeated exposure to dental procedures or clinic visits may evoke psychological trauma, leading to multifaceted negative consequences in the future.

This study aims to compare the effects of an individualized game-based simulation presented through virtual reality (VR) glasses versus the conventional tell-show-do (TSD) technique on children's pain intensity and anxiety during dental procedures.

A total of 88 children, determined through power analysis, aged 6-10 years and attending their first dental visit, will be randomly assigned to two groups using odd-even numbering. The study group (odd numbers) will receive restorative treatment accompanied by a VR-based game, while the other group (even numbers) will undergo treatment using the TSD technique.

In the VR group, children will experience a specially designed interactive game that explains the treatment process step-by-step. The game aims to redirect attention away from discomfort using motivational elements such as visual-auditory stimuli, narrative-driven stages, and the goal of progressing through the game. Behaviors that support cooperation will be embedded as in-game tasks to improve compliance and reduce anxiety.

In the other group, behavior management will be provided using the tell-show-do method. This includes explaining procedures using child-friendly language (tell), demonstrating non-threatening aspects of the instruments and environment (show), and performing the procedures accordingly (do).

After informed consent is obtained, the treating dentist will select teeth based on clinical and radiographic criteria. Dento-alveolar images will be reviewed using VR glasses and explained to the parent, who will also wear VR glasses for an immersive consultation experience. A caries detection tool powered by artificial intelligence will support diagnosis.

Treatments will be performed on the lower primary molars with mesio-occlusal or disto-occlusal caries not involving the pulp.

Pain perception and anxiety will be evaluated using psychometric scales (SCARED, CFSS-DS, Wong-Baker, STAIC) and physiological measurements (pulse oximeter, heart rate) at standardized intervals: before, during, and after treatment.

It is hypothesized that the VR-based game will result in lower anxiety and pain perception, greater cooperation, and more positive dental experiences compared to the tell-show-do method.

DETAILED DESCRIPTION:
Positive experiences during a child's first dental visit contribute to the development of both acute and long-term positive attitudes toward dentists and dental treatments. However, some children may find dental visits stressful or frightening due to several factors, including being in an unfamiliar environment, fear of pain, negative remarks about dentists they might have heard from others, the sounds of dental equipment, bright lights, or even their parents' anxious demeanor. Addressing these fears and implementing strategies to reduce anxiety and alter pain perception can make dental visits smoother. Such measures also positively influence children's oral health, dental development, future dental experiences, eating habits, general health, and self-confidence.

On the contrary, if the first dental experience is associated with pain and anxiety, this can condition children-particularly those who are more sensitive-to develop persistent dental anxiety. In severe cases, repeated exposure to dental procedures or clinic visits may evoke psychological trauma, leading to multifaceted negative consequences in the future.

This study aims to compare the effects of an individualized game-based simulation presented through virtual reality (VR) glasses versus the conventional tell-show-do (TSD) technique on children's pain intensity and anxiety during dental procedures.

A total of 88 children, determined through power analysis, aged 6-10 years and attending their first dental visit, will be randomly assigned to two groups using odd-even numbering. The study group (odd numbers) will receive restorative treatment accompanied by a VR-based game, while the other group (even numbers) will undergo treatment using the TSD technique.

In the VR group, children will experience a specially designed interactive game that explains the treatment process step-by-step. The game aims to redirect attention away from discomfort using motivational elements such as visual-auditory stimuli, narrative-driven stages, and the goal of progressing through the game. Behaviors that support cooperation will be embedded as in-game tasks to improve compliance and reduce anxiety.

In the other group, behavior management will be provided using the tell-show-do method. This includes explaining procedures using child-friendly language (tell), demonstrating non-threatening aspects of the instruments and environment (show), and performing the procedures accordingly (do).

After informed consent is obtained, the treating dentist will select teeth based on clinical and radiographic criteria. Dento-alveolar images will be reviewed using VR glasses and explained to the parent, who will also wear VR glasses for an immersive consultation experience. A caries detection tool powered by artificial intelligence will support diagnosis.

Treatments will be performed on the lower primary molars with mesio-occlusal or disto-occlusal caries not involving the pulp.

To ensure the exclusion of children with underlying psychopathologies, participants will first be screened using the Child Behavior Checklist (CBCL) and the Schedule for Affective Disorders and Schizophrenia for School-Age Children (K-SADS). Only those without psychiatric indications will be included in the study.

Pain perception and anxiety will be evaluated using psychometric scales (SCARED, CFSS-DS, Wong-Baker, STAIC) and physiological measurements (pulse oximeter, heart rate) at four standardized intervals: before treatment, during anesthesia administration, during the procedure, and after treatment.

It is hypothesized that the VR-based game will result in lower anxiety and pain perception, greater cooperation, and more positive dental experiences compared to the tell-show-do method.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6 to 10 years
* No previous dental treatment history
* No systemic or chronic medical conditions
* No mental retardation
* No psychiatric pathology based on CBCL, K-SADS-PL-T, and SCARED (SCARED score <25)
* Presence of dentin caries on mandibular molars (mesio-occlusal or disto-occlusal)
* Signed informed consent by parent/Guardian

Exclusion Criteria:

* Prior dental treatment experience
* SCARED score ≥25
* Diagnosed psychological or developmental disorders
* Acute dental pain or irreversible pulp involvement
* Decline to sign informed consent

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 88 (Estimated)
Dates: Start 2025-09-08 (Actual); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
State-Trait Anxiety Inventory for Children - Dental Version | Time Frame: Baseline (before the treatment) and within 20 minutes after the end of the restorative treatment for each arm.
  Description: A validated self-report questionnaire used to evaluate children's state and trait anxiety levels in dental settings.
  Score Range: 20 to 60 for each subscale (State and Trait). Interpretation: Higher scores indicate greater anxiety levels.
SCARED (Screen for Child Anxiety Related Emotional Disorders) | Time Frame: Baseline (before the treatment) and within 20 minutes after the end of the restorative treatment for each arm.
  Description: A validated self-report tool assessing symptoms of anxiety disorders in children.
  Score Range: 0 to 82. Interpretation: Higher scores reflect greater anxiety. Scores ≥25 suggest clinically significant anxiety.
Pulse Rate Monitoring via Pulse Oximeter | T1: Baseline - before the patient is seated in the dental chair. T2: During local anesthesia administration. T3: During the restorative treatment. T4: Within 5 minutes after completion of the treatment.
  Description: Objective physiological measurement of heart rate used as an indicator of anxiety. Pulse rate will be recorded at multiple standardized time points.
  Score Range: Beats per minute (bpm); continuous numerical data. Interpretation: Higher pulse rates are associated with increased physiological anxiety.
Wong-Baker Faces Pain Rating Scale | Time Frame: After local anesthesia administration and within 20 minutes after the end of the restorative treatment for each arm.
  Description: A self-assessment scale where children rate their pain using illustrated facial expressions.
  Score Range: 0 to 10. Interpretation: Higher scores represent greater perceived pain.
Children's Fear Survey Schedule - Dental Subscale (CFSS-DS) | Time Frame: Within 20 minutes after the end of the restorative treatment for each arm.
  Description: Standardized questionnaire evaluating children's dental-specific fears.
  Score Range: 15 to 75. Interpretation: Higher scores indicate higher dental fear. A score >38 is typically considered high.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara University, Faculty of Dentistry, Pediatric Dentistry Dept, Ankara, Yenimahalle, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie the results reported in the study publication (after deidentification), including raw data for primary and secondary outcome measures, may be shared upon reasonable request. Supporting documentation such as the study protocol and statistical analysis plan may also be made available upon reasonable request.
Supporting Information: Study Protocol, SAP